CLINICAL TRIAL: NCT07177586
Title: A Multicenter, Randomized Controlled Study Comparing the Effectiveness of the New Generation GMA Laryngeal Mask and Conventional Laryngeal Mask in Airway Management During General Anesthesia
Brief Title: New-Generation GMA Laryngeal Mask Airway Versus Conventional Inflatable Laryngeal Mask Airway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: The Second Affiliated Hospital of Zhejiang Chinese Medical University (Other); Red Cross Hospital, Hangzhou, China (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Lanxi People's Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The Second Affiliated Hospital of Jiaxing University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Ruijin Hospital (Other); The Central Hospital of Lishui City (Other); Lishui Country People's Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, xiangming fang, Director, Head of Anesthesiology and Critical Care, Principal Investigator, Professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Laryngeal mask
Record Dates: First submitted 2025-08-29; First posted 2025-09-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Supraglottic Airway Devices Position
Keywords: supraglottic airway device; laryngeal mask

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inflatable LMA Group (Active Comparator): Patients in this group will receive airway management using the standard inflatable LMA (Laryngeal Mask Airway) during general anesthesia. The device will be inserted according to manufacturer guidelines, and sealing pressure, insertion success rate, and ventilation efficacy will be recorded.
  Interventions: Device: Inflatable Laryngeal Mask Airway
- GMA Group (Experimental): Patients in this group will receive airway management using the GMA-Tulip LMA, a modified supraglottic airway device. Insertion technique and outcome measurements (e.g., sealing pressure, ventilation parameters) will be recorded.
  Interventions: Device: GMA Laryngeal Mask Airway

INTERVENTIONS:
Device: GMA Laryngeal Mask Airway — The GMA-Tulip is a new single-use supraglottic airway device (SAD). Device size is selected based on the patient's weight and height, following manufacturer guidelines.
  Other Names: GMA-Tulip LMA
  Arms: GMA Group
Device: Inflatable Laryngeal Mask Airway — The comparator is a conventional inflatable Laryngeal Mask Airway (LMA) of appropriate size (selected by weight/height), inserted using standard clinical protocols.
  Other Names: Cuffed Supraglottic Airway
  Arms: Inflatable LMA Group

SUMMARY:
This study aims to compare the new-generation GMA laryngeal mask airway (LMA) with the traditional inflatable LMA in patients undergoing elective surgery under general anesthesia. The primary objectives are to evaluate the safety, effectiveness, stability, ease of use, and patient comfort of the GMA LMA, providing practical guidance for clinical airway management. Additionally, this research will analyze the anatomical positioning and sealing mechanism of the LMA to identify factors influencing proper alignment and airway sealing. The findings may contribute to future improvements in LMA design, enhancing patient safety and procedural success.

This study is designed for healthcare providers, anesthesiologists, and researchers seeking evidence-based recommendations for LMA selection in clinical practice. Participation involves standard anesthesia procedures with close monitoring to ensure patient safety.

DETAILED DESCRIPTION:
Eligible patients meeting the inclusion criteria were enrolled in the study and randomly assigned into two groups using a random number table: the traditional Inflatable Laryngeal Mask Airway Group (Group L) and the GMA Group (Group G). One day before surgery, the research team conducted preliminary screening of patients scheduled for elective surgery, followed by a preoperative visit to explain the study's purpose, anesthesia considerations, and obtain informed consent. Upon entering the operating room, standard monitoring (ECG, blood pressure, pulse oximetry, etc.) was applied. The research team recorded the patient's actual fasting duration, last intake (food/liquid type), and baseline characteristics, including age, sex, height, weight, BMI, comorbidities, ASA classification, surgical type, and preoperative anxiety level. Airway assessment was reconfirmed. Anesthesia induction was performed with intravenous etomidate, vecuronium, and sufentanil. After loss of consciousness and disappearance of the eyelash reflex, manual ventilation was initiated. Following induction, the laryngeal mask was inserted.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Age 18-75 years;
  2. ASA physical status I-II;
  3. Strict compliance with ASA fasting guidelines;
  4. Normal airway anatomy;
  5. Voluntary participation with signed informed consent.
* Exclusion Criteria:

  1. Pre-existing aspiration risk or gastrointestinal disorders;
  2. Oropharyngeal/laryngeal abnormalities;
  3. Anticipated difficult airway (≥1 of the following):

     BMI >30 kg/m² Mouth opening <3 cm Mallampati class III-IV Restricted neck mobility
  4. Contraindications to LMA use;
  5. Communication or cognitive impairments;
  6. Other exclusions at investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1384 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of anatomical alignment of laryngeal mask | During LMA placement (immediately after insertion)
  Comparison of anatomical positioning success rates between inflatable LMA and GMA-Tulip LMA, assessed by fiberoptic bronchoscopy (FOB).

SECONDARY OUTCOMES:
Sealing pressure and positional stability of the GMA-Tulip versus inflatable LMA | Intraoperative period (from LMA insertion until removal at end of surgery)
  Assess the stability and anti-displacement properties of special body positions (e.g. lateral decubitus, Trendelenburg position) and the laryngeal mask airway under pneumoperitoneum.
First-attempt success rate of LMA | during procedure
  First-attempt success: Successful placement of the laryngeal mask airway on the first attempt without requiring reinsertion
Time to Successful Placement of LMA | during procedure
  Duration (in seconds) from LMA insertion into the oral cavity until final correct positioning is achieved
Hemodynamic response to LMA insertion and removal | Intraoperative period
  Parameters: Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) (measured non-invasively or invasively).
Oxygenation Stability (Intraoperative) | From patient entry into operating room to the time for LMA removal
  Peripheral oxygen saturation (SpO₂) (%) measured by continuous pulse oximetry
Ventilation Parameters (Intraoperative) | from the start of mechanical ventilation after LMA placement to LMA removal
  The measurement of Peak Airway Pressure (Ppeak) in cmH₂O is typically obtained through real-time monitoring by the anesthesia machine's ventilator system.
Feasibility of gastric tube insertion through LMA | During LMA placement (after confirmation of correct LMA position).
  Success rate: Proportion of cases with successful gastric tube placement
LMA-Related Complications | Day 0
  Immediate complications: Visible blood on removal (graded: none/mild/moderate/severe), sore throat , hoarseness, aspiration.
  Pain assessment: NRS for sore throat .
Patient Tolerance Score | Within 60 minutes after LMA removal
  Grade I (Excellent Tolerance) to Grade IV (Severe Intolerance)
Anesthesiologist Satisfaction Survey | Within 30 minutes after surgery completion
  Scale: 1-10 (1 = Very dissatisfied, 10 = Very satisfied)
Surgeon Satisfaction Assessment | Within 30 minutes after surgery completion
  Scale: 1-10 (1 = Very dissatisfied, 10 = Very satisfied)
Patient Satisfaction Survey | Within 24 hours after surgery
  Scale: 1-10 (1 = Very uncomfortable, 10 = Very comfortable)
Ultrasonographic Assessment of Gastric Antrum Cross-Sectional Area (CSA) in Supine Position for Monitoring Gastric Insufflation | Baseline: Within 10 minutes before anesthesia induction; Post-intervention: Within 3 minutes after successful LMA placement; Postoperative: After surgical closure but before LMA removal
  This protocol utilizes point-of-care ultrasound (POCUS) to measure gastric antrum cross-sectional area (CSA) in supine patients, evaluating the risk of perioperative gastric insufflation caused by LMA.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangming Fang, Principal Investigator — Zhejiang University
Locations (1):
- The First affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant confidentiality per institutional policies.

REFERENCES:
- [Background] Zheng J, Du L, Wang J, Zhang L, Chen G. Prewarming i-gel laryngeal mask for mechanical ventilation: a meta-analysis of randomised control trials and trial sequential analysis. BMJ Open. 2021 Aug 10;11(8):e045461. doi: 10.1136/bmjopen-2020-045461. PMID 34376440
- [Background] Luo K, Chen K, Li Y, Ji Y. Clinical evaluation of laryngeal mask airways in video-assisted thoracic surgery: a meta-analysis of randomized controlled trials. J Cardiothorac Surg. 2024 Jun 24;19(1):361. doi: 10.1186/s13019-024-02840-6. PMID 38915035
- [Result] Xu K, Zhang Y, Cui Y, Tian F. Patient-reported outcomes of laryngeal mask anesthesia in thoracoscopic pulmonary wedge resection: A randomized controlled study. Thorac Cancer. 2022 Nov;13(22):3192-3199. doi: 10.1111/1759-7714.14675. Epub 2022 Sep 30. PMID 36178200
- [Result] De Rosa S, Messina A, Sorbello M, Rigobello A, Colombo D, Piccolo A, Bonaldi E, Gennaro P, Urukalo V, Pellizzari A, Bonato R, Carboni SC. Laryngeal Mask Airway Supreme vs. the Spritztube tracheal cannula in anaesthetised adult patients: A randomised controlled trial. Eur J Anaesthesiol. 2019 Dec;36(12):955-962. doi: 10.1097/EJA.0000000000001106. PMID 31644512
- [Result] Wei CF, Chung YT. Laryngeal mask airway facilitates a safe and smooth emergence from anesthesia in patients undergoing craniotomy: a prospective randomized controlled study. BMC Anesthesiol. 2023 Jan 17;23(1):29. doi: 10.1186/s12871-023-01972-x. PMID 36650435